CLINICAL TRIAL: NCT02612623
Title: A Randomized, Parallel, Double-Blind Study to Assess the Efficacy and Tolerability of AF-219 in Subjects With Refractory Chronic Cough
Brief Title: An 8-Week Refractory Chronic Cough Study (MK-7264-021)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Afferent Pharmaceuticals, Inc., a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 7264-021; AF219-021 (Other: Afferent Pharmaceuticals); MK-7264-021 (Other: Merck Protocol Number)
Record Dates: First submitted 2015-11-20; First posted 2015-11-24 (Estimated); Results first posted 2019-11-25 (Actual); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Refractory Chronic Cough
MeSH Terms: conditions — Chronic Cough | interventions — Gefapixant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Gefapixant 15 mg twice daily (Experimental): Two 7.5 mg gefapixant tablets administered by mouth twice daily for 8 weeks
  Interventions: Drug: Gefapixant
- Gefapixant 30 mg twice daily (Experimental): Four 7.5 mg gefapixant tablets administered by mouth twice daily for 8 weeks
  Interventions: Drug: Gefapixant
- Gefapixant 50 mg twice daily (Experimental): One 50 mg gefapixant tablet administered by mouth twice daily for 8 weeks
  Interventions: Drug: Gefapixant
- Placebo to match gefapixant (Experimental): Matching placebo tablets administered by mouth twice daily for 8 weeks
  Interventions: Drug: Placebo (for gefapixant)

INTERVENTIONS:
Drug: Gefapixant — Gefapixant tablets administered by mouth twice daily for 8 weeks
  Other Names: AF-219; MK-7264
  Arms: Gefapixant 15 mg twice daily; Gefapixant 30 mg twice daily; Gefapixant 50 mg twice daily
Drug: Placebo (for gefapixant) — Matching placebo to gefapixant tablets administered by mouth twice daily for 8 weeks
  Arms: Placebo to match gefapixant

SUMMARY:
This was an 8-week randomized, parallel, double-blind, placebo-controlled study of gefapixant (AF-219) in participants with refractory chronic cough.

ELIGIBILITY:
Inclusion Criteria:

* Women and Men between 18 and 80 years of age inclusive
* Have refractory chronic cough
* Women of child-bearing potential must use 2 forms of acceptable birth control
* Have provided written informed consent.
* Are willing and able to comply with all aspects of the protocol.

Exclusion Criteria:

* Current smoker
* Forced Expiratory Volume (FEV1)/Forced Vital Capacity (FVC) < 60%
* History of upper respiratory tract infection or recent significant change in pulmonary status within 4 weeks of the Baseline
* History of opioid use within 1 week of the Baseline Visit
* Body mass index (BMI) <18 kg/m2 or ≥ 40 kg/m2
* History of concurrent malignancy or recurrence of malignancy within 2 years prior to Screening (not including participants with <3 excised basal cell carcinomas)
* Screening systolic blood pressure (SBP) >160 mm Hg or a diastolic blood pressure (DBP) >90 mm Hg
* Significantly abnormal laboratory tests at Screening
* Clinically significant abnormal electrocardiogram (ECG)
* Pregnant or Breastfeeding
* Other severe, acute, or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with trial participation or investigational product administration or may interfere with the interpretation of trial results and, in the judgment of the Investigator or Sponsor, would make the participants inappropriate for entry into this trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-12-17 (Actual); Primary Completion 2016-05-04 (Actual); Study Completion 2016-05-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (10):
- United States (10):
  - Afferent Investigative Site, Mission Viejo, California
  - Afferent Investigative Site, San Jose, California
  - Afferent Investigative Site, Colorado Springs, Colorado
  - Afferent Investigative Site, Largo, Florida
  - Afferent Investigative Site, Charlotte, North Carolina
  - Afferent Investigative Site, Tulsa, Oklahoma
  - Afferent Investigative Site, Dallas, Texas
  - Afferent Investigative Site, San Antonio, Texas
  - Afferent Investigative Site, Bellevue, Washington
  - Afferent Investigative Site, Greenfield, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Male and female participants with treatment-refractory chronic cough were enrolled in this study.
Period: Overall Study
Arm/Group | Gefapixant 15 mg Twice Daily | Gefapixant 30 mg Twice Daily | Gefapixant 50 mg Twice Daily | Placebo to Match Gefapixant
Started (Randomized) | 8 | 6 | 6 | 4
Treated | 8 | 5 | 6 | 4
Completed | 7 | 5 | 5 | 4
Not Completed | 1 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants who had received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Gefapixant 15 mg Twice Daily | Gefapixant 30 mg Twice Daily | Gefapixant 50 mg Twice Daily | Placebo to Match Gefapixant | Total
Number analyzed (Participants) | 8 | 5 | 6 | 4 | 23
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.30 (10.39) | 66.60 (7.30) | 62.70 (11.04) | 63.50 (2.38) | 62.80 (8.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 4 | 5 | 3 | 20
  Male | 0 | 1 | 1 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 8 | 5 | 6 | 3 | 22
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 8 | 5 | 5 | 4 | 22
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Cough Frequency [Mean (Standard Deviation); unit: Coughs/hour] — Cough monitoring was conducted for 24 hours while awake, at pre-dose on Day 0. The cough frequency is the coughs/hr over the 24 hour period. An independent cough monitoring core lab provided documentation of the time of each cough event over each 24-hour period. Population: All randomized participants who took at least 1 dose of study medication and provided at least one baseline and at least one post-dose observation.
  Coughs/hour
    number analyzed (Participants) | 7 | 5 | 5 | 4 | 21
    (all) | 57.6 (35.98) | 42.7 (21.22) | 41.0 (29.98) | 60.4 (38.84) | 50.6 (30.98)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Awake Cough Frequency After 8 Weeks of Treatment.
Description: Cough monitoring was conducted for 24 hours while awake, at pre-dose on Day 0, and after administration of the study drug on Day 56. The cough frequency is the coughs/hr over each 24 hour period. An independent cough monitoring core lab provided documentation of the time of each cough event over each 24-hour period. A negative change indicates a decrease in cough frequency, while a positive change indicates an increase in cough frequency.
Time Frame: Baseline and Week 8 (Day 56)
Population: All randomized participants who took at least 1 dose of study medication and provided at least one baseline and at least one post-dose observation.
Measure: Mean (Standard Deviation); unit: Coughs/hour
Arm/Group | Gefapixant 15 mg Twice Daily | Gefapixant 30 mg Twice Daily | Gefapixant 50 mg Twice Daily | Placebo to Match Gefapixant
Number analyzed (Participants) | 7 | 5 | 5 | 4
Coughs/hour | -7.5 (40.58) | -16.9 (13.68) | -18.5 (26.88) | 0.3 (24.96)
Statistical Analysis 1: Comparison: Gefapixant 15 mg Twice Daily vs Placebo to Match Gefapixant; Least squares mean (LSM) difference: Mixed effect repeated measures model (MMRM) uses the change from baseline as the dependent variable, and includes the treatment group, visit day, and the interaction between treatment and visit as fixed factors, and baseline as a covariate; Test type: Other; LSM Difference = -0.56, 95% CI 2-sided [-2.08 to 0.96] — Gefapixant minus Placebo
Statistical Analysis 2: Comparison: Gefapixant 30 mg Twice Daily vs Placebo to Match Gefapixant; LSM difference: MMRM uses the change from baseline as the dependent variable, and includes the treatment group, visit day, and the interaction between treatment and visit as fixed factors, and baseline as a covariate; Test type: Other; LSM Difference = -0.71, 95% CI 2-sided [-2.34 to 0.92] — Gefapixant minus Placebo
Statistical Analysis 3: Comparison: Gefapixant 50 mg Twice Daily vs Placebo to Match Gefapixant; [analysis description as in outcome 1, analysis 2]; Test type: Other; LSM Difference = -1.35, 95% CI 2-sided [-2.99 to 0.30] — Gefapixant minus Placebo
Statistical Analysis 4: Comparison: Gefapixant 15 mg Twice Daily vs Placebo to Match Gefapixant; Estimated Percentage Change: MMRM uses the change from baseline as the dependent variable, and includes the treatment group, visit day, and the interaction between treatment and visit as fixed factors, and baseline as a covariate; Test type: Other; Percentage Change = -42.6, 95% CI 2-sided [-87.5 to 162.3] — 100 x [(Exponent of LSM Difference) minus 1]
Statistical Analysis 5: Comparison: Gefapixant 30 mg Twice Daily vs Placebo to Match Gefapixant; [analysis description as in outcome 1, analysis 4]; Test type: Other; Percentage Change = -50.8, 95% CI 2-sided [-90.3 to 151.1] — 100 x [(Exponent of LSM Difference) minus 1]
Statistical Analysis 6: Comparison: Gefapixant 50 mg Twice Daily vs Placebo to Match Gefapixant; [analysis description as in outcome 1, analysis 4]; Test type: Other; Percentage Change = -74.0, 95% CI 2-sided [-95.0 to 34.7] — 100 x [(Exponent of LSM Difference) minus 1]

ADVERSE EVENTS:
Time Frame: Up to 14 days after Day 57 (up to 71 days)
Description: The population analyzed was all randomized participants who had received at least 1 dose of study drug.
Groups:
- Placebo: Matching placebo tablets administered by mouth twice daily for 8 weeks
- Gefapixant 15 mg: Two 7.5 mg gefapixant tablets administered by mouth twice daily for 8 weeks
- Gefapixant 30 mg: Four 7.5 mg gefapixant tablets administered by mouth twice daily for 8 weeks
- Gefapixant 50 mg: One 50 mg gefapixant tablet administered by mouth twice daily for 8 weeks
Arm/Group | Placebo | Gefapixant 15 mg | Gefapixant 30 mg | Gefapixant 50 mg
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/8 | 0/5 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/8 | 1/5 | 0/6
Other Adverse Events (participants affected / at risk) | 4/4 | 5/8 | 4/5 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=4) | Gefapixant 15 mg (N=8) | Gefapixant 30 mg (N=5) | Gefapixant 50 mg (N=6)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=4) | Gefapixant 15 mg (N=8) | Gefapixant 30 mg (N=5) | Gefapixant 50 mg (N=6)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia oral (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Inflammation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tinea pedis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Stress fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 2 (2) | 2 (2) | 4 (5)
Hypogeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results obtained during the course of this study will be kept confidential and will not be disclosed in whole or in part to others or used for any purpose other than reviewing or performing the study without the written consent of the Sponsor. No data collected as part of this study will be utilized in any written work, including publications, without the written consent of the Sponsor.